CLINICAL TRIAL: NCT07169227
Title: The Comparison of the Efficacy of Lidocaine, Paracetamol, and Dexmedetomidine in Preventing Rocuronium Injection Pain
Brief Title: Lidocaine, Paracetamol, and Dexmedetomidine for Rocuronium Injection Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Sibel Catalca, principal investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KA25/209
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Propofol Injection Pain; Rocuronium Injection Pain
Keywords: lidocaine; dexmedetomidine; paracetamol
MeSH Terms: interventions — Dexmedetomidine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine (Active Comparator): Patients who were administered lidocaine before anesthesia induction.
  Interventions: Drug: Lidocaine %2 ampoule
- Paracetamol (Experimental): Patients who were administered paracetamol before anesthesia induction.
  Interventions: Drug: paracetamol
- Dexmedetomidine (Experimental): Patients who were administered dexmedetomidine before anesthesia induction.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Lidocaine %2 ampoule — Patients who were administered 40 mg lidocaine.
  Arms: Lidocaine
Drug: Dexmedetomidine — Patients who were administered 0.25 mg/kg dexmedetomidine.
  Arms: Dexmedetomidine
Drug: paracetamol — Patients who were administered 50 mg paracetamol.
  Arms: Paracetamol

SUMMARY:
Propofol and rocuronium may cause pain during intravenous injection. Various pharmacological agents are used to reduce the incidence and severity of injection pain. Among the most commonly used agents for this purpose are lidocaine, various opioids, ketamine, paracetamol, and dexmedetomidine. The aim of this study was to evaluate the comparative effect of intravenous dexmedetomidine and paracetamol versus lidocaine in preventing propofol- and rocuronium-induced pain during anesthesia induction.

DETAILED DESCRIPTION:
General anesthesia induction is initiated with propofol, and after loss of consciousness is achieved, rocuronium is administered to provide muscle relaxation. Propofol and rocuronium may cause pain during intravenous injection, with an incidence ranging from 20% to 100% for propofol and from 22% to 84% for rocuronium. The current hypothesis regarding the mechanism of pain associated with intravenous drug injection is that stimulation of polymodal nociceptors triggers the release of endogenous pain mediators such as prostaglandins. This stimulation is thought to be related to the non-physiological osmolarity or pH of the drug solution.

The pain that occurs during anesthesia induction may lead to undesirable reflex movements, which can result in accidental dislodgement of the intravenous catheter. In addition, in response to strong nociceptive stimulation, it may also contribute to the development of increased arterial blood pressure and tachycardia. Various pharmacological and non-pharmacological strategies have been investigated to reduce the incidence and severity of injection pain. Among the most commonly used agents for this purpose are lidocaine, various opioids, magnesium, sodium bicarbonate, ketamine, paracetamol, and dexmedetomidine.

Although lidocaine is frequently used to prevent propofol/rocuronium injection pain during anesthesia, propofol or rocuronium pain can still occur in up to 30% of cases, even with lidocaine administration. Therefore, there is currently no pharmacological agent in the literature that has been definitively confirmed to reduce propofol/rocuronium pain.

Paracetamol is a widely used agent for pain management and as an antipyretic, although its precise molecular mechanism of action is not fully understood. However, the antinociceptive effects of paracetamol are thought to occur through both peripheral and central mechanisms via inhibition of cyclooxygenase-2 (COX-2). With its peripheral effects, paracetamol is thought to reduce propofol- and rocuronium-induced injection pain and the associated involuntary withdrawal movements . In addition, paracetamol has been shown to selectively suppress peripheral PGE₂ release and to increase COX-2 gene expression in an acute inflammation model. Another study reported that paracetamol exhibits selectivity in inhibiting the synthesis of prostaglandins and related factors. Furthermore, although paracetamol does not inhibit COX enzymes at therapeutic concentrations in vitro, it has been reported to inhibit a variant of COX enzymes in vivo.

Dexmedetomidine is an α₂-adrenergic receptor agonist with supraspinal, spinal, and peripheral effects, possessing strong sedative, analgesic, and sympatholytic properties. Alpha-2 receptors are found in blood vessels and inhibit the release of norepinephrine. Although some studies in the literature have reported that dexmedetomidine reduces propofol- and rocuronium-induced pain, there are also studies that do not support this finding. Moreover, the effective optimal dose of this agent has not yet been clearly established.

The aim of this study was to evaluate the comparative effect of intravenous dexmedetomidine and paracetamol versus lidocaine in preventing propofol- and rocuronium-induced pain during anesthesia induction.

The goal of this study is to identify an effective pharmacological agent to reduce propofol and rocuronium injection pain. This study is a prospective, randomised study involving 170 subjects and they will assessed on the incidence and severity of rocuronium and propofol pain during anesthesia induction. Outcomes from this study can be extended to patients who will be receiving general anaesthesia tube to reduce the incidence and severity of propofol and rocuronium injection pain.

ELIGIBILITY:
Inclusion Criteria:

Patients who will receive propofol and rocuronium 18 - 65 years No psychiatric disorders Elective surgery Those who accept the research No history of allergy to any of the drugs used in the study Patients in American Society of Anesthesiologists (ASA) I and II class

Exclusion Criteria:

Patients with chronic pain syndromes Patients with difficult intravenous access Patients with advanced heart block or heart failure Patients with uncontrolled hypertension (Systolic blood pressure >160 mmHg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Rocuronium Withdrawal Movement Score | Immediately after rocuronium injection
  Score evaluating involuntary withdrawal movements in response to rocuronium injection (0 = No movement, 1 = Movement only at the wrist, 2 = Movement involving the upper arm and shoulder of the injected arm, 3 = Widespread movement in multiple extremities or full-body withdrawal)

SECONDARY OUTCOMES:
Propofol Pain Score | Immediately after propofol injection
  Score assessing the intensity of pain during propofol injection. ıt will be assessed with 11-point Visual Analog Scale (0: No pain at all, 10: Worst pain imaginable in my life).

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Çatalca, Dr., Principal Investigator — Baskent University, Adana Dr. Turgut Noyan Hospital
Locations (1):
- Baskent University, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uzun S, Erden IA, Canbay O, Aypar U. The effect of intravenous paracetamol for the prevention of rocuronium injection pain. Kaohsiung J Med Sci. 2014 Nov;30(11):566-9. doi: 10.1016/j.kjms.2014.08.002. Epub 2014 Sep 22. PMID 25458046
- [Background] He L, Xu JM, He T, Liu L, Zhu R. Dexmedetomidine pretreatment alleviates propofol injection pain. Ups J Med Sci. 2014 Nov;119(4):338-42. doi: 10.3109/03009734.2014.941049. Epub 2014 Oct 24. PMID 25342205
- [Background] Kwak HJ, Kim JY, Kim YB, Min SK, Moon BK, Kim JY. Pharmacological prevention of rocuronium-induced injection pain or withdrawal movements: a meta-analysis. J Anesth. 2013 Oct;27(5):742-9. doi: 10.1007/s00540-013-1595-7. Epub 2013 Mar 22. PMID 23519582